# This is the consent form & assent script for the study entitled

"Retrieval-Based Word Learning in Developmental Language Disorder"

No NCT number has been assigned yet

6/7/2023

### RESEARCH PARTICIPANT CONSENT FORM

# Retrieval-based Word Learning Principal Investigator: Laurence B. Leonard, PhD Department of Speech, Language, & Hearing Sciences Purdue University

### **Key Information**

Please take time to review this information carefully. This is a research study. Your child's participation in this study is voluntary which means that you or your child may choose not to have your child participate at any time without penalty or loss of benefits to which you are otherwise entitled. You may ask questions of the researchers about the study whenever you would like. If you decide to have your child take part in the study, you will be asked to sign this form. Be sure you understand what you will do and any possible risks or benefits. The purpose of this study is to understand how children learn new words. The duration of the study will be 1 session to determine if your child is eligible. These sessions will last approximately 60 minutes each. If your child qualifies, there will be an additional 5 sessions that will each last approximately 60 minutes.

### What is the purpose of this study?

You are being asked to participate in this study so that we can examine how children learn new words. We would like to enroll 274 children in this study.

# What will I do if I choose to be in this study?

We will ask your child to participate in a variety of activities. These involve looking at pictures and listening to sentences presented on a computer. Novel words will be used to label pictures of plants and animals. Your child will respond by pointing to pictures and by using the novel words to label pictures. Your child will also watch videos in which characters do novel actions described by novel verbs. He/she will then be prompted to describe actions using the novel verbs. In addition, some standardized tests of language, speech and cognitive abilities will be administered in order to obtain more information about your child. All sessions will be audiorecorded and/or videorecorded.

### How long will I be in the study?

The research activities will be conducted at in our lab at Purdue University in 6 one-hour sessions. Over the course of the study, there will be two points at which sessions will be scheduled on consecutive days. Otherwise, sessions will be scheduled weekly at mutually convenient times. Each of the periods will be broken up into smaller segments to prevent fatigue and boredom.

# What are the possible risks or discomforts?

There is risk of breach of confidentiality. However, safeguards are in place to minimize this risk, as outlined in the Confidentiality section. The activities that your child will participate in do not have any more risks than what he/she would encounter in everyday activities. In-person research carries with it the risk of contracting COVID-19. However, precautions will be taken to minimize this risk at all times. Specifically, research staff will strictly adhere to all guidelines for PPE and cleaning outlined in the Protect Purdue guidelines. You may choose to have your child wear a mask, but s/he will be asked to remove it for short periods to record verbal responses.

### Are there any potential benefits?

There are no direct benefits to your child of the research activities. The research activities are not intended for diagnosis or treatment purposes. However, after your child's participation is complete, we will provide you with a report, summarizing test scores and other information about your child that we gained during the research activities.

### Will I receive payment or other incentive?

| The receive payment of other meentives | |
|---|---|
| Your child will be tested in 1 session to determine if he/she meets the criteria which determine el | igibility to participate |
| in this study. If your child does not qualify, you will be paid \$10.00 for each of the testing session | ns as compensation |
| | (continued on p.2) |

| Parent Initials | Date | Researcher Initials | Date |
|-----------------|------|---------------------|------|
| Parent Initials | Date | | |

for your expenses in bringing the child to the testing site and your child will receive a small toy after each session. If your child does qualify, you will be paid \$10.00 for each of the testing sessions and will be offered the opportunity to continue participation in the research project. If you choose to have your child continue, you will be paid \$10.00 for each of the remaining 5 1-hour research periods and your child will receive a small toy after each session. There is no compensation for your child's participation in the therapy and play activities (and no fee is charged).

# Will information about me and my participation be kept confidential?

This project is funded by the National Institutes of Health (NIH). The project's research records may be reviewed by departments at the Purdue University responsible for research oversight, or the NIH, to ensure those participants' rights are being protected. All of the research activities will be audio- and/or videorecorded to ensure the accuracy of our transcription of your child's responses. The identity of all participants will remain confidential. Data for those children deemed ineligible for the study will be destroyed immediately. Children who participate in the study will be assigned a participant identification number; all records, data, and publications will contain only this ID number. All data will be stored, using the same identification system, in file cabinets in a locked laboratory in Lyles-Porter Hall (rooms 3132, 3172, 3182) or on password protected computers. The participant ID key will be separated from the data in a locked file cabinet in LPH 3182. The data will be used in the present research project and will be archived for use in future associated projects. Three years after all related publications are completed, the data and participant ID key will be destroyed. Paper data will be shredded and electronic records erased. Only the research team directly involved with the project will have access to the data. In order for us to compensate you for your expenses using a Purdue-issued check, we will submit your name, social security number and address to the business office of Purdue University using a secure file sharing system.

This study meets the NIH definition of a Clinical Trial. As such, a description of this clinical trial will be available on ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the Website will include a summary of the results. You can search this Website at any time.

Sometimes it is helpful for us to be able to play audio-or videorecordings of children when we discuss our research in the classroom or at professional meetings. In such cases, we ensure that the child's name is not used on the recording. Place an "X" on the line below that indicates your preference regarding the use of audio- and/or videorecordings for this purpose.

| this purpose. | y p |
|---|---|
| I voluntarily give my c<br>I do not give my conse | consent for audio- and/or videorecordings of my child to be used. ent for audio- and/or videorecordings of my child to be used. Parent Initials |
| information about the study so that you can | you about future studies in our lab. When we contact you, we would provide decide whether or not you want your child to participate. You may, at any acted. Place an "X" on the line below if interested: ct me about future studies. |
| Certificate of Confidentiality | |
| with this Certificate may not disclose or use<br>federal, state, or local civil, criminal, admir<br>evidence, for example, if there is a court su<br>biospecimens protected by this Certificate of | f Confidentiality from the National Institutes of Health. The researchers information, documents, or biospecimens that may identify you in any distrative, legislative, or other action, suit, or proceeding, or be used as become, unless you have consented for this use. Information, documents, or cannot be disclosed to anyone else who is not connected with the research with the required disclosure (such as to report shill always or company is called |
| * ' | w that requires disclosure (such as to report child abuse or communicable ivil, criminal, administrative, legislative, or other proceedings, see below); |
| if you have consented to the disclosure, inc | luding for your medical treatment; or if it is used for other scientific protecting research subjects. For additional information about CoCs see |

| Parent Initials | Date | Researcher Initials | Date _ |
|-----------------|------|---------------------|--------|
| Parent Initials | Date | | |

# What are my rights if I take part in this study?

You do not have to participate in this research project. If you do agree to participate you can withdraw your participation at any time without penalty. At each session, we will ask your child for his/her verbal consent to participate (e.g., "Do you want to play the listening game today?"). If your child does not give consent, the activity will be suspended until a later time. If at any time during a research activity, your child gives verbal or non-verbal indication of a refusal to continue, the activity will be suspended until a later time.

# Who can I contact if I have question about the study?

If you have any questions, comments, or concerns about this research project, you can talk to one of the researchers: P.I. Dr. Laurence B. Leonard, at (765) 494-3794 or Pat Deevy at (765)496-1821, <a href="mailto:deevy@purdue.edu">deevy@purdue.edu</a>. If you have questions about your rights while taking part in the study or have concerns about the treatment of research participants, contact the Human Research Protection Program (HRPP) at Purdue University at (765) 494-5942, <a href="mailto:irb@purdue.edu">irb@purdue.edu</a> or write to HRPP, Ernest C. Young Hall, 10th Floor-Room 1032, 155 S. Grant Street, West Lafayette, IN 47907-2114.

# **Documentation of Informed Consent**

I have had the opportunity to read this consent from and have the research study explained. I have had the opportunity to ask questions about the research study, and my questions have been answered. I am prepared to participate in the research study described above. I will receive a copy of this consent form after I sign it.

| Parent/Legal Guardian's Signature | Date |
|-----------------------------------|------|
| Parent/Legal Guardian's Name | |
| Parent/Legal Guardian's Signature | Date |
| Parent/Legal Guardian's Name | |
| Child Participant's Name | |
| Researcher's Signature | Date |